CLINICAL TRIAL: NCT06194214
Title: A Phase I, Open-label, Fixed-sequence, Drug Interaction Study to Investigate the Effect of Single and Multiple Oral Doses of LOXO-305 on the Pharmacokinetics of Multiple Oral Doses of Digoxin (P-Glycoprotein Substrate) in Healthy Subjects
Brief Title: A Drug Drug Interaction (DDI) Study of Pirtobrutinib (LOXO-305) and Digoxin (P-Glycoprotein Substrate) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20021; J2N-OX-JZNT (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-13; First posted 2024-01-08 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — pirtobrutinib; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Digoxin + Pirtobrutinib (Experimental): Participants received oral dose of
  * 0.25 mg digoxin twice daily (BID) on Day 1
  * 0.25 mg digoxin once daily (QD) from Day 2 to Day 7
  * 200 mg Pirtobrutinib in combination with 0.25 mg digoxin QD starting from Day 8 to Day 16
  Interventions: Drug: Pirtobrutinib; Drug: Digoxin

INTERVENTIONS:
Drug: Pirtobrutinib — Administered Orally.
  Other Names: LOXO-305; LY3527727
Drug: Digoxin — Administered Orally.

SUMMARY:
The main purpose of this study is to evaluate the effect of Pirtobrutinib (LOXO-305) on multiple oral doses of digoxin (P-gp substrate) when administered as single and multiple doses by collecting the blood samples and conducting the blood tests to measure how much digoxin is in the bloodstream and how the body handles and eliminates it in healthy participants. The study will also evaluate the safety and tolerability of Pirtobrutinib. Participants will stay in this study for up to 58 days, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive
* Male and female participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods
* Must have comply with all study procedures, including the 20-night stay at the Clinical Research Unit (CRU) and follow-up phone call

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Positive serologic test for hepatitis B surface antigen (HBsAg), hepatitis B virus immunoglobulin M (HBV IgM) core antibody, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening
* Positive polymerase chain reaction (PCR) test for COVID-19 at Screening or Check-in (Day -1)
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee)
* Have previously completed or withdrawn from any other study investigating Pirtobrutinib (LOXO-305) and have previously received the investigational product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Digoxin + Pirtobrutinib
Started | 16
Received at Least 1 Dose of Study Drug | 16 (* Received at least 1 dose of Digoxin alone; N=16 * Received at least 1 dose of Pirtobrutinib in combination with Digoxin; N=16)
Completed | 15
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve From Hour 0 to the Last Measurable Concentration (AUC[0-t]) of Digoxin in Plasma
Description: PK: AUC[0-t] of Digoxin was reported.
Time Frame: Day 7 and Day 8: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours postdose; Day 16: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours postdose
Population: All enrolled population who had received at least one dose of digoxin had at least one quantifiable PK concentration and for whom at least one PK parameter was computed. Number analyzed refer to participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
hour*nanogram per milliliter (h*ng/mL)
  Day 7 | 14.6 (21.1)
  Day 8 | 17.1 (19.6)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 48.9 (22.0)

2. Primary Outcome: PK: Area Under the Concentration During a Dosing Interval (AUC [Tau]) of Digoxin in Plasma
Description: PK: AUC [tau] of Digoxin was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
h*ng/mL
  Day 7 | 14.7 (21.1)
  Day 8 | 17.2 (19.6)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 20.4 (23.4)

3. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Digoxin in Plasma
Description: PK: CL/F of Digoxin in plasma was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour(L/h)
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
liter per hour(L/h)
  Day 7 | 17.0 (21.1)
  Day 8 | 14.5 (19.6)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 12.2 (23.4)

4. Primary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of Digoxin in Plasma
Description: PK: Cmax of Digoxin was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
nanogram per milliliter (ng/mL)
  Day 7 | 1.57 (26.1)
  Day 8 | 2.38 (27.7)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 2.45 (42.0)

5. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Digoxin in Plasma
Description: PK: Tmax of Digoxin was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
hour
  Day 7 | 1.27 [0.750 to 3.00]
  Day 8 | 1.25 [0.750 to 3.00]
  Day 16: number analyzed (Participants) | 15
  Day 16 | 1.00 [0.750 to 2.50]

6. Primary Outcome: PK: Mean Residence Time (MRT) of Digoxin in Plasma
Description: PK: MRT of Digoxin was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
hours
  Day 7 | 52.2 (49.1)
  Day 8 | 65.2 (47.2)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 60.4 (52.5)

7. Primary Outcome: PK: Cumulative Amount of Drug Excreted Unchanged in Urine (Ae) of Digoxin
Description: PK: Ae of Digoxin in urine was reported. The urine sampling time points from pre-dose through 24 hours post-dose were used to assess this outcome.
Time Frame: Day 7 and Day 16: Predose, 6, 12, 24 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
mg
  Day 7 | 0.123 (23.3)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 0.148 (18.2)

8. Primary Outcome: PK: Fraction of Digoxin Excreted Unchanged in Urine (Fe) Expressed as Percentage of Dose Excreted
Description: PK: Fe of Digoxin was reported. The urine sampling time points from pre-dose through 24 hours post-dose were used to assess this outcome.
Time Frame: Day 7 and Day 16: Predose, 6, 12, 24 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose excreted in urine
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
percentage of dose excreted in urine
  Day 7 | 49.2 (23.3)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 59.4 (18.2)

9. Primary Outcome: PK: Renal Clearance (CLr) of Digoxin in Plasma
Description: PK: CLr of Digoxin in plasma was reported.
Time Frame: Day 7: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours postdose; Day 16: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
L/h
  Day 7 | 8.35 (15.0)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 7.28 (17.0)

10. Primary Outcome: PK: Area Under the Concentration From Hour 0 to the Last Measurable Concentration (AUC0-t) of Pirtobrutinib in Plasma
Description: PK: AUC[0-t] of Pirtobrutinib was reported.
Time Frame: Day 8: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours postdose; Day 16: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours postdose
Population: All enrolled population who had received at least one dose of Pirtobrutinib had at least one quantifiable PK concentration and for whom at least one PK parameter was computed. Number analyzed refer to participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
h*ng/mL
  Day 8 | 48400 (16.3)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 189000 (25.8)

11. Primary Outcome: PK: Area Under the Concentration During a Dosing Interval (AUCtau) of Pirtobrutinib in Plasma
Description: PK: AUCtau of Pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
h*ng/mL
  Day 8 | 48600 (16.3)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 106000 (21.0)

12. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Pirtobrutinib in Plasma
Description: PK: CL/F of Pirtobrutinib in plasma was reported.
Time Frame: Day 16: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours postdose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 15
L/h | 1.89 (21.0)

13. Primary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of Pirtobrutinib in Plasma
Description: PK: Cmax of Pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
ng/mL
  Day 8 | 4330 (17.1)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 7530 (17.9)

14. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Pirtobrutinib in Plasma
Description: PK: Tmax of Pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
hours
  Day 8 | 2.50 [1.00 to 3.00]
  Day 16: number analyzed (Participants) | 15
  Day 16 | 2.50 [0.500 to 4.00]

15. Primary Outcome: PK: Mean Residence Time (MRT) of Pirtobrutinib in Plasma
Description: PK: MRT of Pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Digoxin + Pirtobrutinib
Number analyzed (Participants) | 16
hours
  Day 8 | 22.6 (18.7)
  Day 16: number analyzed (Participants) | 15
  Day 16 | 30.5 (17.5)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 27
Description: All participants who had received at least 1 dose of study drug. The adverse events were analyzed and reported according to the study treatment pre-specified in the statistical analysis plan.
Groups:
- 0.25 mg Digoxin: * Participants who received 0.25 mg digoxin orally BID on Day 1.
  * Participants who received 0.25 mg digoxin orally QD from Day 2 to Day 7.
- 200 mg Pirtobrutinib + 0.25 mg Digoxin: * Participants who received 200 mg Pirtobrutinib in combination with 0.25 mg digoxin QD starting from Day 8 to Day 16.
Arm/Group | 0.25 mg Digoxin | 200 mg Pirtobrutinib + 0.25 mg Digoxin
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 5/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.25 mg Digoxin (N=16) | 200 mg Pirtobrutinib + 0.25 mg Digoxin (N=16)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Medical device site erythema (General disorders) | 2 (2) | 0 (0)
Medical device site injury (General disorders) | 1 (1) | 0 (0)
Medical device site pruritus (General disorders) | 1 (1) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT06194214/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT06194214/SAP_001.pdf